CLINICAL TRIAL: NCT01928628
Title: A Randomized, Multicenter, Parallel Design Phase III Clinical Study to Evaluate the Efficacy and Safety of the Combination of Lercanidipine/Valsartan in Hypertensive Patients Who Are Not Adequately Controlled on Lercanidipine 10mg Monotherapy.
Brief Title: Phase III Clinical Study to Evaluate the Efficacy and Safety of the Combination of Lercanidipine/Valsartan in Hypertensive Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LG-ZVCL005
Record Dates: First submitted 2013-08-21; First posted 2013-08-27 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-08

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — lercanidipine; Valsartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lercanidipine 10mg (Active Comparator): 1 Tablet of Zanidip ® 10mg + 1 Tablet of L10/V80 Placebo + 1 Tablet of L10/V160 Placebo (8wks)
  Interventions: Drug: Lercanidipine 10mg; Drug: Lercanidipine10mg /Valsartan 80mg Placebo; Drug: Lercanidipine 10mg /Valsartan 160mg Placebo
- Lercanidipine10mg /Valsartan 80mg (Experimental): 1 Tablet of Zanidip ® 10mg Placebo +1 Tablet of L10/V80 + 1 Tablet of L10/V160 Placebo (8wks)
  Interventions: Drug: Lercanidipine10mg /Valsartan 80mg; Drug: Lercanidipin 10mg Placebo; Drug: Lercanidipine 10mg /Valsartan 160mg Placebo
- Lercanidipine 10mg /Valsartan 160mg (Experimental): 1 Tablet of Zanidip ® 10mg Placebo + 1 Tablet of L10/V80 Placebo + 1 Tablet of L10/ V160 (8wks)
  Interventions: Drug: Lercanidipine 10mg /Valsartan 160mg; Drug: Lercanidipin 10mg Placebo; Drug: Lercanidipine10mg /Valsartan 80mg Placebo

INTERVENTIONS:
Drug: Lercanidipine 10mg
  Arms: Lercanidipine 10mg
Drug: Lercanidipine10mg /Valsartan 80mg
  Arms: Lercanidipine10mg /Valsartan 80mg
Drug: Lercanidipine 10mg /Valsartan 160mg
  Arms: Lercanidipine 10mg /Valsartan 160mg
Drug: Lercanidipin 10mg Placebo
  Arms: Lercanidipine 10mg /Valsartan 160mg; Lercanidipine10mg /Valsartan 80mg
Drug: Lercanidipine10mg /Valsartan 80mg Placebo
  Arms: Lercanidipine 10mg; Lercanidipine 10mg /Valsartan 160mg
Drug: Lercanidipine 10mg /Valsartan 160mg Placebo
  Arms: Lercanidipine 10mg; Lercanidipine10mg /Valsartan 80mg

SUMMARY:
This study aims to compare and assess the efficacy and the safety of the combination agent of Lercanidipine and Valsartan and monotherapy of Lercanidipine alone in patients with essential hypertension

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 20 to ≤75 years old
* Patient with essential hypertension

Exclusion Criteria:

* When the BP level measured at screening was sitDBP>120 mmHg or sitSBP >180 mmHg
* Patient with difference in repeatedly measured blood pressures from the selected arm at screening was sitSBP≥ 20mmHg or sitDBP ≥ 10mmHg

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 449 (Actual)
Dates: Start 2012-05; Primary Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Change in mean sitDBP from week 0 to week 40 | 40 weeks

SECONDARY OUTCOMES:
Response rate at week 4 and 8 | 4 weeks and 8 weeks
  Proportion (%) of patients with mean sitDBP<90mmHg or proportion (%) of patients with mean reduction of sitDBP ≥10mmHg from week 0

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Na SH, Lee HY, Hong Baek S, Jeon HK, Kang JH, Kim YN, Park CG, Ryu JK, Rhee MY, Kim MH, Hong TJ, Choi DJ, Cho SW, Cha DH, Jeon ES, Kim JJ, Shin JH, Park SH, Lee SH, John SH, Shin ES, Kim NH, Lee SY, Kwan J, Jeong MH, Kim SW, Jeong JO, Kim DW, Lee NH, Park WJ, Ahn JC, Won KH, Uk Lee S, Cho JH, Kim SK, Ahn T, Hong S, Yoo SY, Kim SY, Kim BS, Juhn JH, Kim SY, Lee YJ, Oh BH. Evaluation of the Efficacy and Safety of the Lercanidipine/Valsartan Combination in Korean Patients With Essential Hypertension Not Adequately Controlled With Lercanidipine Monotherapy: A Randomized, Multicenter, Parallel Design, Phase III Clinical Trial. Clin Ther. 2015 Aug;37(8):1726-39. doi: 10.1016/j.clinthera.2015.05.512. Epub 2015 Jul 8. PMID 26164786